CLINICAL TRIAL: NCT06573463
Title: Longevity of Prefabricated Band and Loop Versus Conventional Band and Loop Space Maintainers in Children With Prematurely Lost First Primary Molars
Brief Title: Longevity of Prefabricated Band and Loop Versus Conventional Band and Loop Space Maintainers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lamis Abdelkhalek Mohamed Badawi, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Conventional vs prefabricated
Record Dates: First submitted 2024-08-16; First posted 2024-08-27 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Premature Tooth Exfoliation

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial, parallel group, allocation ratio 1:1 Framework superiority
Who Masked: Outcomes Assessor
Masking Description: Blinding will not be feasible neither for the operator nor the patient. As there are some differences in the clinical steps, the form of the appliances and number of needed visits.
  Outcome assessor and Statistician will be blinded from the intervention and control not knowing which group represents which procedure.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional band and loop (Active Comparator): Conventional band and loop is the most widely used space maintainer, and the most effective. It shows high success rate and good patient compliance, but it needs more than one visit to be applied.
  Interventions: Device: Conventional Band and loop
- Prefabricated band and loop (Active Comparator): Prefabricated space maintainer requires only one visit as it fits into the patient's mouth at the clinic without needing the dental lab. It comes in a kit with different band sizes.
  Interventions: Device: Prefabricated band and loop

INTERVENTIONS:
Device: Prefabricated band and loop — Prefabricated space maintainer requires only one visit as it fits into the patient's mouth at the clinic without needing the dental lab. It comes in a kit with different band sizes.
  Other Names: Ready-made band and loop; Chairside band and loop
  Arms: Prefabricated band and loop
Device: Conventional Band and loop — Conventional band and loop is the most widely used space maintainer, It shows high success rate and good patient compliance, but needs more than one visit due to the laboratory work.
  Arms: Conventional band and loop

SUMMARY:
To assess the longevity of prefabricated versus conventional band and loop space maintainers in children with prematurely lost first primary molars.

A Randomized Clinical Trial

DETAILED DESCRIPTION:
When considering gingival health and cement dissolution, does the longevity of the prefabricated band and loop differ from the conventional band and loop constructed following the premature loss of the lower first primary molars?

The concept of preserving space after premature tooth loss has been recognized for over a century. Conventional appliances are used successfully as space maintainers, but some disadvantages like the need for at least two visits to deliver the appliance due to laboratory work, will definitely affect its role during the general anesthesia.

The prefabricated space maintainer requires only one visit as it is fitted into the patient's mouth at the clinic without needing the dental lab. This provides a good impact on apprehensive children as it reduces the number of visits and chairside time. Prefabricated space maintainers could be a new alternative to the conventional fixed space maintainers used in pediatric dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Patients having mandibular first deciduous molar indicated for extraction due to extensive coronal caries beyond possible repair, root caries and/or failed pulp therapy.
* Caries free, or restored mandibular second primary molars and deciduous canines on the side of the extraction maintained throughout the entire follow-up period.
* Children are classified as cooperative or potentially cooperative according to Wright's classification of child behavior.
* According to space analysis, available space is less than or equal to the needed space
* 1/3 to less than 2/3 of the root of the permanent successor is formed to the prematurely lost primary molars
* Children are mentally capable of communication.
* Children aged 4-6 years

Exclusion Criteria:

* Children with any parafunctional habits.
* Children with previous allergies to stainless steel.
* Permanent successors with 2/3 of its roots formed and space analysis does not indicate the fabrication of space maintainer.
* Parental refusal of participation.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Gingival Health | 3 month and 9 month
  By using gingival index of Loe and Silness ,scores gingival inflammation from 0-3
  0 = normal gingiva
  1. = mild inflammation: slight change in color, slight edema, no bleeding on probing
  2. = moderate inflammation: redness, edema, glazing, or bleeding on probing
  3. = severe inflammation: marked redness and edema, tendency toward spontaneous bleeding
Cement integrity | 3 month and 9 month
  Visual inspection of cement solution by using blunt periodontal explorer and mirror, Binary (Yes, No)

SECONDARY OUTCOMES:
Space loss between the abutment teeth. | 0 month and 9 month
  Change in distance measured on digital cast between the mesial midpoint of the second deciduous molar and the distal midpoint of the primary canine in mm.
Change in arch dimension: | 0 month and 9 month
  1. Arch perimeter: Measured on digital cast as a sum of the incisor, canine and molar segment widths in mm.
  2. Inter canine width : Measured on digital cast from cusp tip of canine on one side to cusp tip of canine on the other side in mm.
  3. Intermolar width: Measured on a digital cast from central fossa of the second primary molar on one side to central fossa of the second primary molar on the other side in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Y El Kharadly, Lecturer, Study Director — October 6 University
Locations (1):
- Cairo university, Cairo, Egypt

REFERENCES:
- [Background] Kamki H, Kalaskar R, Balasubramanian S, Badhe H, Kalaskar A. Clinical Effectiveness of Fiber-reinforced Composite Space Maintainer and Band and Loop Space Maintainer in a Pediatric Patient: A Systematic Review and Meta-analysis. Int J Clin Pediatr Dent. 2021;14(Suppl 1):S82-S93. doi: 10.5005/jp-journals-10005-2044. PMID 35082473
- [Background] Tahririan D, Safaripour M, Eshghi A, Bonyadian AH. Comparison of the longevity of prefabricated and conventional band and loops in children's primary teeth. Dent Res J (Isfahan). 2019 Nov 12;16(6):428-434. eCollection 2019 Nov-Dec. PMID 31803390
- [Background] Padma Kumari B, Retnakumari N. Loss of space and changes in the dental arch after premature loss of the lower primary molar: a longitudinal study. J Indian Soc Pedod Prev Dent. 2006 Jun;24(2):90-6. doi: 10.4103/0970-4388.26023. PMID 16823234
- [Background] Thakur B, Bhardwaj A, Luke AM, Wahjuningrum DA. Effectiveness of traditional band and loop space maintainer vs 3D-printed space maintainer following the loss of primary teeth: a randomized clinical trial. Sci Rep. 2024 Jun 18;14(1):14081. doi: 10.1038/s41598-024-61743-7. PMID 38890410
- [Background] Zhao J, Jin H, Li X, Qin X. Dental arch spatial changes after premature loss of first primary molars: a systematic review and meta-analysis of split-mouth studies. BMC Oral Health. 2023 Jun 28;23(1):430. doi: 10.1186/s12903-023-03111-x. PMID 37380944